CLINICAL TRIAL: NCT02905942
Title: A Single Center Randomized Controlled Trial of the Efficacy and Safety of PEG-rhG-CSF After Autologous Hematopoietic Stem Cell Transplantation for Lymphoma Patients
Brief Title: PEG-rhG-CSF in Lymphoma Patients After Autologous Hematopoietic Stem Cell Transplantation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Jun Zhu, Director, Peking University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-JYL-20150830
Record Dates: First submitted 2016-09-14; First posted 2016-09-19 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-09

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — pegylated granulocyte colony-stimulating factor

ARMS (2):
- PEG-rhG-CSF (Experimental): Patients in PEG-rhG-CSF group received PEG-rhG-CSF day +1 after transplantation.
  Interventions: Drug: PEG-rhG-CSF
- rhG-CSF (Active Comparator): Patients in control group received rhG-CSF day +1 after transplantation.
  Interventions: Drug: rhG-CSF

INTERVENTIONS:
Drug: PEG-rhG-CSF — PEG-rhG-CSF was given day +1 after autologous stem cell transplantation with a dose of 100μg/kg(bw).For patients more than 45kg, 6mg was suggested.
  Arms: PEG-rhG-CSF
Drug: rhG-CSF — rhG-CSF was given day +1 after transplantation with a dose of 5μg/kg once per day
  Arms: rhG-CSF

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of PEG-rhG-CSF on the recovery of hematopoietic function after autologous stem cell transplantation in patients with lymphoma.

DETAILED DESCRIPTION:
At present, there is few related research of Recombinant Human Granulocyte Colony-stimulating Factor applying to AHSCT in China. The purpose of the study is to evaluate the efficacy and safety of PEG-rhG-CSF in lymphoma patients after autologous hematopoietic stem cell transplantation. Eligible patients were randomly assigned to PEG-rhG-CSF group or rhG-CSF group. Patients in PEG-rhG-CSF group received PEG-rhG-CSF day +1 after transplantation with a dose of 100μg/kg. Patients with the weight more than 45kg were suggested a dose of 6 mg. Patients in control group received rhG-CSF day +1 after transplantation with a dose of 5μg/kg once per day until the recovery of neutrophil.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with age between 18 and 65 years.
2. Lymphoma patients with the requirement for autologous hematopoietic stem cell transplantation.
3. The collected CD34+ cells≥1×10E6/kg.
4. ECOG score ≤2.
5. Heart and lung is normal.
6. Blood creatinine ≤1.5×ULN.
7. ALT, AST, TBIL ≤2 ×ULN
8. Not in pregnancy.
9. Written informed consent are acquired.

Exclusion Criteria:

1. Had received autologous hematopoietic stem cell transplantation or allogeneic transplantation.
2. Severe or uncontrolled infectious diseases: HIV, HCV, syphilis, ALT, chronic hepatitis B.
3. Serious complications, such as severe infection, heart, lung, liver and kidney dysfunction.
4. LVEF <55%.
5. Allergic to the product or other biological products from genetically engineered Escherichia coli strains.
6. Refused to take contraceptive measures during the study period and the subsequent 1 years.
7. Severe mental or neurological disorders.
8. Serious heart, lung, central nervous system disorders.
9. Sickle cell anemia, hemolytic anemia and other hematologic diseases.
10. Participate in other drugs clinical trials 30 days before the screening.
11. Other situation that investigators consider as contra-indication for this study.

    -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2015-12; Primary Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Time to neutrophil engraftment | 30days

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhu, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital, Beijing, China